CLINICAL TRIAL: NCT04215263
Title: Risk Factors of Post Operative Cognitive Dysfunction (POCD) in General Anesthesia Patients Underwent Noncardiac and Non Neurological Procedures.
Brief Title: Risk Factors of POCD in General Anesthesia Patients Underwent Noncardiac and Non Neurological Procedures.
Status: Completed | Type: Observational
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Aries Perdana, Principal Investigator, Indonesia University
Other Study IDs: IndonesiaUAnes 044
Record Dates: First submitted 2019-12-30; First posted 2020-01-02 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Undergoing General Anaesthesia
Keywords: postoperative cognitive dysfunction; geriatrics; general anaesthesia
MeSH Terms: conditions — Postoperative Cognitive Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Geriatric patient underwent general anesthesia procedure: geriatric patients (≥60 years) ware assessed for cognitive impairment after general anesthesia for non-neurologic noncardiac surgery.
  Interventions: Other: Questionaire

INTERVENTIONS:
Other: Questionaire — Patient was assessed using mini international neuropsychiatric interview

SUMMARY:
The study was a prospective cohort study to assess the effect of age, duration of anesthesia, repeated surgery, and type of surgery on cognitive impairment in 108 geriatric patients (≥60 years) who underwent general anesthesia for non-neurologic noncardiac surgery.

DETAILED DESCRIPTION:
The study was a prospective cohort study, assessing the effect of age, duration of anesthesia, repeated surgery, and type of surgery on cognitive impairment in 108 geriatric patients (≥60 years) who underwent general anesthesia for non-neurologic noncardiac surgery. The study used cognitive tests such as RAVLT, TMT, and Digit span tests. POCD definition is reduction in postoperative cognitive function by as much as 20% at a minimum of 2 cognitive tests.

ELIGIBILITY:
Inclusion Criteria:

* geriatric patient (age over 60) underwent noncardiac non-neurological procedure under general anesthesia
* patient can do reading and writing
* patient can speak in Bahasa
* signing informed consent

Exclusion Criteria:

* patient with cognitive impairment or psychiatric disorder such as delirium, amnesia, anxiety disorder, or depression.
* patient under psychotropic drugs or narcotics.
* patient with history of brain tumor, head injury or motoric disturbance and disability that can disturbed neurocognitive test

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Geriatric patient (age over 60) underwent noncardiac non-neurological procedure under general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-07-05 (Actual); Study Completion 2019-07-05 (Actual)

PRIMARY OUTCOMES:
Mini International Neuropsychiatric Interview | 7 days
  Score was assessed using 6 forms

CONTACTS AND LOCATIONS:
Overall Officials: Aries Perdana, MD, Principal Investigator — Indonesia University
Locations (1):
- Indonesia University, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] BEDFORD PD. Adverse cerebral effects of anaesthesia on old people. Lancet. 1955 Aug 6;269(6884):259-63. doi: 10.1016/s0140-6736(55)92689-1. No abstract available. PMID 13243706
- [Result] Strom C, Rasmussen LS, Sieber FE. Should general anaesthesia be avoided in the elderly? Anaesthesia. 2014 Jan;69 Suppl 1(Suppl 1):35-44. doi: 10.1111/anae.12493. PMID 24303859
- [Result] Rundshagen I. Postoperative cognitive dysfunction. Dtsch Arztebl Int. 2014 Feb 21;111(8):119-25. doi: 10.3238/arztebl.2014.0119. PMID 24622758
- [Result] Canet J, Raeder J, Rasmussen LS, Enlund M, Kuipers HM, Hanning CD, Jolles J, Korttila K, Siersma VD, Dodds C, Abildstrom H, Sneyd JR, Vila P, Johnson T, Munoz Corsini L, Silverstein JH, Nielsen IK, Moller JT; ISPOCD2 investigators. Cognitive dysfunction after minor surgery in the elderly. Acta Anaesthesiol Scand. 2003 Nov;47(10):1204-10. doi: 10.1046/j.1399-6576.2003.00238.x. PMID 14616316
- [Result] van Harten AE, Scheeren TW, Absalom AR. A review of postoperative cognitive dysfunction and neuroinflammation associated with cardiac surgery and anaesthesia. Anaesthesia. 2012 Mar;67(3):280-93. doi: 10.1111/j.1365-2044.2011.07008.x. PMID 22321085